CLINICAL TRIAL: NCT01915524
Title: An Exploratory, Open-label Phase Ib Study of RNActive®-Derived Cancer Vaccine and Local Radiation as Consolidation and Maintenance Treatment in Patients With Stage IV NSCLC and a Response or Stable Disease After First-line Chemotherapy or Therapy With an EGFR Tyrosine Kinase Inhibitor
Brief Title: Trial of RNActive®-Derived Cancer Vaccine and Local Radiation in in Stage IV Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment in stratum 3: enrolled only 2 instead of 8 pts. within predicted time
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-9202-006
Record Dates: First submitted 2013-07-18; First posted 2013-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CV9202 and local radiation (Experimental): CV9202 consisting of 6 RNActive-derived molecules coding for 6 different NSCLC associated antigens.
  local radiation (4x5 Gy)
  Interventions: Biological: CV9202; Radiation: local radiation

INTERVENTIONS:
Biological: CV9202 — Intradermal injection of CV9202
Radiation: local radiation — Radiotherapy will be administered in 4 daily fractions of 5 GY each to be administered within one week

SUMMARY:
The purpose of this study is to determine whether the new RNActive derived lung cancer vaccine CV9202 in combination with local radiation therapy is safe, tolerable and immunogenic for the consolidation and maintenance treatment of stage IV non small cell lung cancer (NSCLC) after first-line chemotherapy or therapy with an EGFR tyrosine kinase inhibitor.

DETAILED DESCRIPTION:
The Phase Ib study is the first clinical study with the new lung cancer vaccine CV9202. The vaccine is composed of 6 RNActive compounts, each encoding for a different antigen which is overexpressed in NSCLC compared to healthy tissue.

In order to enhance the immunogenic effect of the cancer vaccine, the study treatment will include local radiation (4 x 5 Gy), which is a well-established palliative radiation regimen that can be safely applied to metastatic lesions in the lung, bone, and soft tissue, and is well tolerated.

Patients will be enrolled into 3 strata based on histologic and molecular subtypes as follows:

Stratum 1: Patients with metastatic stage IV NSCLC and non-squamous histology, without activating epidermal growth factor receptor (EGFR) mutations, who have achieved partial response (PR) or stable disease (SD) after at least 4 cycles of platinum- and pemetrexed-based first-line chemotherapy, and an indication for maintenance therapy with pemetrexed.

Stratum 2: Patients with stage IV NSCLC and squamous cell histology, who achieved PR or SD after at least 4 cycles of platinum-based and non-platinum compound first-line chemotherapy.

Stratum 3: Patients with stage IV NSCLC and non-squamous histology, harboring an activating EGFR mutation, who have achieved PR after up to 6 months or SD after 3 - 6 months of treatment with an EGFR TKI.

In each patient, the vaccine will be administered until progression and the need to start a subsequent systemic second-line treatment, or occurrence of unacceptable toxicity requiring treatment discontinuation, whichever comes first.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients >= 18 years of age with histologically or cytologically-confirmed stage IV NSCLC, and a confirmed EGFR mutation status in case of non-squamous cell histology

   * Stratum 1: Non-squamous NSCLC without activating EGFR mutation
   * Stratum 2: Squamous NSCLC
   * Stratum 3: Non-squamous NSCLC harboring an activating EGFR mutation
2. PR or SD according to RECIST Version 1.1 after first-line therapy which should have consisted of:

   * Stratum 1: PR or SD after cisplatin or carboplatin and pemetrexed treatment (at least 4 cycles)
   * Stratum 2: PR or SD after cisplatin or carboplatin and a non-platinum compound treatment (at least 4 cycles)
   * Stratum 3: PR after up to 6 months or SD after at least 3 and up to 6 months of gefitinib or erlotinib treatment
3. For patients in stratum 1, maintenance therapy with pemetrexed should be indicated as to the investigator's opinion
4. Presence of at least one tumor lesion that is eligible for radiation with 4 x 5 GY, and at least one additional measurable tumor lesion according to RECIST Version 1.1.

   Tumor lesions eligible for radiation are:
   * Bone metastases
   * Lymph nodes in the paraclavicular, axillary or cervical regions
   * Skin or subcutaneous metastases
   * For patients in strata 1 and 2 only: Thoracic lesions (centrally located lung tumor, lymph nodes in the lung hilus or mediastinum)
5. Performance Status: Eastern Cooperative Oncology Group (ECOG) 0 to 1

Key Exclusion Criteria:

1. Previous active immunotherapy for NSCLC (including vaccination, therapy with anti-CTLA4 antibodies)
2. Estimated life expectancy ≤ 3 months
3. Need for immunosuppressive treatment including daily systemic steroid doses of ≥ 10 mg prednisone equivalent per day
4. Active skin disease (e.g. atopic dermatitis) in the areas for vaccine injection (upper arms or thighs) not allowing intradermal injections into areas of healthy skin
5. Concurrent or planned major surgery
6. Prior splenectomy or prior allogeneic bone marrow transplantation
7. History of pneumonitis
8. Documented history or active autoimmune disorders with the exception of vitiligo, diabetes mellitus type 1 or autoimmune thyroiditis requiring hormone replacement only
9. Primary or secondary immune deficiency
10. Allergies to any components of the study drug including allergy to protamine hydrochloride (e.g. allergy to protamine-containing insulin) or fish allergy
11. Seropositive for HIV, HBV, HCV or any other infection requiring anti-infection therapy
12. For patients in stratum 3: persisting >= grade 3 skin rash at time of enrollment
13. Known brain metastases with the exception of stable metastases being treated with stereotactic radiation or surgery)

    **Local German Amendment: 13. Brain metastases (symptomatic or asymptomatic) or leptomeningeal involvement
14. Uncontrolled medical condition considered as high risk for the treatment with an investigational drug (e.g. unstable diabetes mellitus, vena-cava-syndrome, uncontrolled pleural effusion, pericardial effusion, symptomatic congestive heart failure (New York Heart Association 3 or 4), unstable angina pectoris/myocardial infarction within the previous 6 months, significant cardiac arrhythmia, history of stroke or transient ischemic attack within the previous 6 months, severe hypertension according to WHO criteria, and uncontrolled systolic blood pressure ≥ 180 mmHg at the time of enrollment
15. For patients planned to undergo radiation of thoracic lesions: inadequate lung function dependent on the intended tumor volume and location to be irradiated (to be assessed by the radio oncologist)
16. History of encephalitis or multiple sclerosis
17. Active inflammatory conditions such as inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related >= grade 3 adverse events (AEs). | up to 40 months
  Events are graded by the investigator using the NCI CTCAE Scale (version 4.0) which provides a grading scale for each AE term. Grade 3 = Severe Grade 4 = Life-threatening or disabling
  Interim safety evaluations will be performed:
  * After treatment and observation of the first 6 patients until Day 43 in a given stratum.
    - If >= 2 out of 6 patients experience treatment-related >= grade 3 AEs, enrollment in that stratum will be suspended.
  * After the first 6 patients (enrolled in stratum 1 or 2) have received radiation of thoracic lesions and have been monitored for toxicity until Day 57:
    * If >= 2 out of 6 patients experience >= grade 3 radiation pneumonitis, radiation of thoracic lesions will be suspended for further patients.
    * For strata 1 and 2, CV9202 administration and radiation of thoracic lesions will be considered safe for further evaluation if ≤ 20% of patients experience a >= grade 3 radiation pneumonitis and no patients experience grade 4 radiation pneumonitis.

SECONDARY OUTCOMES:
humoral and cellular immune responses against the 6 antigens encoded by CV9202. | assessments at baseline, Day 19, Day 61 after start of study treatment
broadening of humoral immune responses (antigen spreading, i.e. change in serum antibody patterns) against a panel of tumor antigens not covered by the vaccine. | Assessment at baseline, Day 19, Day 61 and 12 weeks, 24 weeks and 48 weeks after Day 57
overall tumor response. | At Screening and every 6 weeks during study treatment until progression up to 18 months after start of treatment of the last patient enrolled
progression free survival (PFS) and time to start of second-line treatment | every 6 weeks up to 18 months after start of treatment of the last patient enrolled
response to second-line cancer treatment | every 3 months after completion of study treatment until death, withdrawal of informed consent, or loss to follow-up or until up to 18 months after start of treatment of the last patient enrolled
overall survival (OS) from time of first vaccination. | From first study treatment until time of death assessed up to 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Zippelius, Prof. Dr., Principal Investigator — University Hospital Basel, Clinic for Medical Oncology
Locations (13):
- Innsbruck Medical University, Department of Internal Medicine V (Hematology and Oncology), Innsbruck, Austria
- Germany (8):
  - HELIOS Klinikum Emil von Behring GmbH, Berlin
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Kliniken der Stadt Köln gGmbH, Cologne
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - University Hospital Frankfurt, Department of Medicine II: Hematology/Oncology, Frankfurt
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - University Medical Center Mainz, III. Medical Clinic and Policlinic, Mainz
  - Pius-Hospital Oldenburg, Oldenburg
- Switzerland (4):
  - University Hospital Basel, Clinic for Oncology, Basel
  - Kantonsspital Graubünden, Chur
  - Kantonspital St. Gallen, Sankt Gallen
  - Kantonspital Winterthur, Oncology, Winterthur

REFERENCES:
- [Derived] Papachristofilou A, Hipp MM, Klinkhardt U, Fruh M, Sebastian M, Weiss C, Pless M, Cathomas R, Hilbe W, Pall G, Wehler T, Alt J, Bischoff H, Geissler M, Griesinger F, Kallen KJ, Fotin-Mleczek M, Schroder A, Scheel B, Muth A, Seibel T, Stosnach C, Doener F, Hong HS, Koch SD, Gnad-Vogt U, Zippelius A. Phase Ib evaluation of a self-adjuvanted protamine formulated mRNA-based active cancer immunotherapy, BI1361849 (CV9202), combined with local radiation treatment in patients with stage IV non-small cell lung cancer. J Immunother Cancer. 2019 Feb 8;7(1):38. doi: 10.1186/s40425-019-0520-5. PMID 30736848
- [Derived] Sebastian M, Papachristofilou A, Weiss C, Fruh M, Cathomas R, Hilbe W, Wehler T, Rippin G, Koch SD, Scheel B, Fotin-Mleczek M, Heidenreich R, Kallen KJ, Gnad-Vogt U, Zippelius A. Phase Ib study evaluating a self-adjuvanted mRNA cancer vaccine (RNActive(R)) combined with local radiation as consolidation and maintenance treatment for patients with stage IV non-small cell lung cancer. BMC Cancer. 2014 Oct 6;14:748. doi: 10.1186/1471-2407-14-748. PMID 25288198
- See also: Click here for more information about CureVac — http://www.curevac.de